CLINICAL TRIAL: NCT02902250
Title: The Comparative Study About the Effect of Vertebral Body Decompression Procedure and Conservative Treatment for Benign Vertebral Compression Fracture - Prospective Randomized Control Study
Brief Title: The Comparative Study About the Effect of Vertebral Body Decompression Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Decon_001
Record Dates: First submitted 2016-09-10; First posted 2016-09-15 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Osteoporotic Vertebral Compression Fracture
Keywords: Vertebroplasty; Core decompression; Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Decompression; Conservative Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompression (Experimental): bone marrow decompression at fractured vertebral body
  Interventions: Procedure: Decompression
- Conservative Treatment (Active Comparator): Conservative Treatment for compression fracture
  Interventions: Procedure: Conservative Treatment

INTERVENTIONS:
Procedure: Decompression — vertebral body decompression in compression fracture
  Arms: Decompression
Procedure: Conservative Treatment — Conservative Treatment in vertebral compression fracture
  Arms: Conservative Treatment

SUMMARY:
The purpose of this study is to compare the treatment efficacy between vertebral body decompression procedure and conservative treatment with non-inferiority design

ELIGIBILITY:
Inclusion Criteria:

* osteoporotic vertebral compression fracture

Exclusion Criteria:

* malignancy or inflammatory disease
* severe pain in other joints
* coagulopathy
* an inappropriate person considered by investigator

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | until 3 months after procedure
  Pain status

SECONDARY OUTCOMES:
Oswestry Disability Index | until 3 months after procedure
  Health status
EQ5D-5L | until 3 months after procedure
  Quality of Life
Leed Dyspepsia Questionnaire | until 3 months after procedure
  Abdominal discomfort d/t medication and injection
Radiographic outcome | until 3 months after procedure
  Compression rate

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Min Park, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyounggido, South Korea

IPD SHARING:
Plan to Share IPD: Undecided